CLINICAL TRIAL: NCT05371613
Title: A Phase 2/3, Multicenter, Double-Blind, Randomized Study to Determine the Efficacy and Safety of Tividenofusp Alfa (DNL310) vs Idursulfase in Pediatric and Young Adult Participants With Neuronopathic or Non-Neuronopathic Mucopolysaccharidosis Type II
Brief Title: A Study to Determine the Efficacy and Safety of Tividenofusp Alfa (DNL310) vs Idursulfase in Pediatric and Young Adult Participants With Neuronopathic (nMPS II) or Non-Neuronopathic Mucopolysaccharidosis Type II (nnMPS II)
Acronym: COMPASS
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNLI-E-0007; 2024-510990-21-00 (EU CTIS Number); 2021-005200-35 (EudraCT Number)
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Mucopolysaccharidosis II
Keywords: Hunter Syndrome; MPS II; nMPS II; nnMPS II
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death | interventions — idursulfase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A: Participants with nMPS II (Experimental)
  Interventions: Drug: tividenofusp alfa; Drug: idursulfase
- Cohort B: Participants with nnMPS II (Experimental)
  Interventions: Drug: tividenofusp alfa; Drug: idursulfase
- Open-label Treatment Phase (Experimental): Participants who meet pre-specified criteria may receive DNL310 or idursulfase
  Interventions: Drug: tividenofusp alfa; Drug: idursulfase

INTERVENTIONS:
Drug: tividenofusp alfa — Intravenous repeating dose
Drug: idursulfase — Intravenous repeating dose

SUMMARY:
This is a Phase 2/3, multiregional, two-arm, double-blind, randomized, active (standard-of-care)-controlled study of the efficacy and safety of tividenofusp alfa (DNL310), an investigational central nervous system (CNS)-penetrant enzyme-replacement therapy (ERT) for mucopolysaccharidosis type II (MPS II).

Participants may also qualify to enter an open-label treatment phase with DNL310 or idursulfase based on pre-specified criteria.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants aged ≥2 to <6 years (Cohort A) or ≥6 to <26 years (Cohort B)
* Confirmed diagnosis of MPS II (for Cohort A, nMPS II; for Cohort B, nnMPS II)
* Have no history of treatment with enzyme replacement therapy (ERT) OR not have received continuous ERT for 4 months prior to screening OR be on maintenance ERT and have tolerated idursulfase for a minimum of 4 months prior to screening

Key Exclusion Criteria:

* Have a documented mutation of other genes or genetic diagnosis accounting for developmental delay
* Previously received an iduronate 2-sulfatase (IDS) gene therapy or stem cell therapy
* Received any CNS-targeted MPS ERT within 6 months prior to screening
* Have a contraindication for lumbar punctures and/or magnetic resonance imaging (MRI)
* Participated in any other investigational drug study or used an investigational drug within 60 days prior to screening or intend to receive another investigational drug during the study

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in cerebrospinal fluid (CSF) heparan sulfate (HS) concentration (Cohort A) | 24 weeks
Change from baseline in the Vineland Adaptive Behavior Scale, Third Edition (Vineland-3)(Cohort A) | 96 weeks

SECONDARY OUTCOMES:
Change from baseline in the Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III)(Cohort A only) | 96 weeks
Change from baseline in the Vineland-3 Adaptive Behavior Composite (ABC; Cohort A only) | 96 weeks
Change from baseline in serum neurofilament light chain (NfL) (Cohort A only) | 96 weeks
Change from baseline in distance walked in the Six-Minute Walk Test (6MWT; Cohort B only) | 48 weeks
Percent change from baseline in the sum of urine HS and dermatan sulfate (DS) concentrations (Cohorts A and B) | up to 48 weeks
Liver volume within the normal range (normal vs abnormal) as measured by magnetic resonance imaging (MRI) (Cohorts A and B) | 48 weeks
Spleen volume within the normal range (normal vs abnormal) as measured by MRI (Cohorts A and B) | 48 weeks
Improvement in Parent/Caregiver Global Impression of Change (CaGI-C) Overall MPS II (Cohorts A and B) | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jose Alcantara Rodriguez, PharmD, Study Director — Denali Therapeutics Inc.
Locations (32):
- United States (8):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Ann and Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Hackensack University Medical Center, Hackensack, New Jersey
  - UNC Children's Research Institute, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The University of Texas Medical School at Houston, Houston, Texas
  - University of Utah, PPDS, Salt Lake City, Utah
- Sanatorio Mater Dei, Buenos Aires, Argentina
- Women's and Children's Hospital, North Adelaide, Australia
- Belgium (2):
  - UZ Antwerpen, Antwerp, Antwerpen
  - Universitair Ziekenhuis Brussel, Jette, Brussels Capital
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre (HCPA) - PPDS, Porto Alegre
  - Instituto Fernandes Figueira, Rio de Janeiro
- Canada (3):
  - University of Alberta - Faculty of Medicine & Dentistry, Edmonton, Alberta
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
- Vseobecna Fakultni Nemocnice V Praze, Prague, Czechia
- Hôpital Jeanne de Flandre, Lille, France
- Germany (2):
  - SphinCS, Höchheim, Hochheim
  - Medizinische Universität Lausitz - Carl Thiem, Cottbus
- Azienda Sanitaria Universitaria Friuli Centrale - PO Universitario Santa Maria della Misericordia, Udine, Italy
- Erasmus Medical Center - Sophia Children's Hospital, Rotterdam, Rotterdam, Netherlands
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona, Barcelona
  - Hospital Infantil Universitario Niño Jesus, Madrid, Madrid
- Drottning Silvias Barn Och Ungdomssjukhus, Gothenburg, Sweden
- Turkey (Türkiye) (2):
  - Cukurova University Medical Faculty Balcali Hospital, Adana
  - Gazi Universitesi Tip Fakultesi, Çankaya
- United Kingdom (4):
  - Great Ormond Street Hospital for Children, London, London
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - Royal Free Hospital, London
  - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Denali Therapeutics — https://www.denalitherapeutics.com/